CLINICAL TRIAL: NCT00067886
Title: Matrix Metalloproteinases and Diabetic Nephropathy
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK62999; R01DK062999 (NIH)
Record Dates: First submitted 2003-08-29; First posted 2003-09-01 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 1; Diabetic Nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Matrix metalloproteinases (MMPs) are a family of protein-degrading enzymes that are involved in the breakdown and remodeling of many tissues and organs. Abnormal activity of these enzymes has been implicated in many disease processes including rheumatoid arthritis, dental disease and metastatic cancer. Recent studies also suggest that elevations in blood sugar may abnormally effect MMP enzyme activity. Decreased activity of some of these MMP enzymes may be a partial cause of the abnormal enlargement of the kidney (renal hypertrophy) seen at the start of diabetic kidney disease (nephropathy). Preliminary clinical data from our laboratory confirm that children with newly diagnosed type 1 diabetes mellitus (DM) have lower blood levels of some of these enzymes at the time of very high blood sugar readings. However, these enzyme levels become normal again as blood sugar levels improve with insulin treatment. In the present study, we propose to investigate the hypothesis that MMPs are involved in the cause of diabetic kidney disease by measuring concentrations of specific MMPs and some related proteins in the blood and urine of patients with type 1 DM who are between the ages of 14-40 years. We will enroll some patients who are recently diagnosed with diabetes, some who have had diabetes for several years, but without signs of kidney disease, and some with long-term diabetes and various degrees of kidney disease. Continuous Subcutaneous Glucose Monitoring, conducted for 3-4 days, will also be provided as a part of this study, to determine how different levels of blood sugar control might relate to different levels of MMP enzyme activity in the blood. We anticipate that this study will help to establish a link between abnormal MMP activity and the cause of nephropathy in type 1 DM, allowing scientists to design better therapies for the prevention and treatment of diabetes-related kidney problems.

ELIGIBILITY:
Type 1 Diabetes with or without kidney disease and past puberty.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Type 1 Diabetes mellitus, ages 14-40 years.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2003-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Thrailkill, MD, Principal Investigator — Arkansas Chilldren's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital/University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Thrailkill KM, Bunn RC, Moreau CS, Cockrell GE, Simpson PM, Coleman HN, Frindik JP, Kemp SF, Fowlkes JL. Matrix metalloproteinase-2 dysregulation in type 1 diabetes. Diabetes Care. 2007 Sep;30(9):2321-6. doi: 10.2337/dc07-0162. Epub 2007 Jun 11. PMID 17563344